CLINICAL TRIAL: NCT06399367
Title: Investigation of Lipedema, Lymphedema and Vascular Malformations by Multispectral Optoacoustic Tomography (MSOT)
Status: Enrolling by invitation | Type: Observational
Sponsor: University Hospital Goettingen (Other)
Responsible Party: Principal Investigator, Laura Hansen, Laura Hansen, Resident Physician, Department of Plastic and Reconstructive Surgery, University Hospital Goettingen
Other Study IDs: 16/10/19
Record Dates: First submitted 2024-02-02; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Lipedema; Lymphedema; Vascular Malformations
MeSH Terms: conditions — Lipedema; Lymphedema; Vascular Malformations

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Lipedema/MSOT Cohort: MSOT measurements are carried out on 50 subjects with changes in the subcutaneous fatty tissue (e.g. lipedema). In these studies, adult patients (>18 years, <80 years) are included with the indicators mentioned below, after risk information and voluntary consent.
  1. Typical tenderness in the calf, back of the knee or lateral thigh
  2. Tendency to hematoma in areas affected by edema
  3. Typical appearance of fatty tissue distribution with dent formation, asymmetry in lateral comparison and increased circumference
  4. Tendency to edema throughout the day with typical feeling of pressure/pain
  5. Unsuccessful conservative therapy attempts and weight loss attempts
  Interventions: Diagnostic Test: MSOT
- Non-Lipedem/MSOT Cohort: MSOT measurements are carried out on 50 subjects with clinically healthy subcutaneous fatty tissue. In these studies, adult patients (>18 years, <80 years) are included after exclusion of the indicators mentioned below, after risk information and voluntary consent.
  1. Typical tenderness in the calf, back of the knee or lateral thigh
  2. Tendency to hematoma in areas affected by edema
  3. Typical appearance of fatty tissue distribution with dent formation, asymmetry in lateral comparison and increased circumference
  4. Tendency to edema throughout the day with typical feeling of pressure/pain
  5. Unsuccessful conservative therapy attempts and weight loss attempts.
  Interventions: Diagnostic Test: MSOT

INTERVENTIONS:
Diagnostic Test: MSOT — The MSOT system used consists of a laser in the visible near-infrared and far-infrared wavelength range (660nm-1300nm) and an ultrasonic sensor connected to a computer. Using optical components, the area to be measured is illuminated with ultra-short light pulses of selectable wavelength. The light is absorbed to varying degrees inside the object - depending on the properties of the tissue. The absorption of light leads to local microscopic volume fluctuations and thereby emits pressure waves in the ultrasonic range (photoacoustic effect). MSOT enables non-invasive, non-ionizing 2D imaging with high spatial resolution (80 μm), which enables specific visualization of endogenous tissue pigments such as collagen fibers, fat, melanin, oxyhemoglobin and deoxyhemoglobin.

SUMMARY:
This study aims to analyze the fatty tissue architecture of the subcutaneous tissue in patients from the plastic surgery department.

Plastic surgery patients show a wide variety of subcutaneous fatty tissue structures during clinical examination. These include patients with edema of the extremities such as lipedema or lymphedema.

Fatty tissue architecture plays a major role in our everyday lives, as wound healing and scar formation, for example, are influenced by the blood flow to the overlying skin. The fatty tissue architecture, especially in the subcutaneous fatty tissue, also plays a major role in our appearance. An analysis of the architecture can potentially provide information about the genesis of different skin fold formations. The aim of this study is to quantitatively describe structural differences in adipose tissue architecture.

Adipose tissue architecture is still a largely unexplored area because imaging has not been possible to date. MSOT imaging is similar to conventional sonography in that a transducer is placed on the skin and energy is supplied to the tissue by pulsed laser light instead of sound. On a macroscopic level, this leads to a constant change of minimal oscillations of individual tissue components. The resulting sound waves can then be detected by the same transducer. Previous studies have shown that the quantitative determination of hemoglobin can be used to obtain information on blood circulation and inflammatory activity. In the extended spectrum, in contrast, not only hemoglobin and its oxygenation stages but also other biomarkers such as collagens and lipids can be detected. This is very useful for imaging of fat, lymphatics and normal and abnormal blood vessels in vascular malformations.

This process was largely researched by the working group of Prof. Ntziachristos (Helmholtz Center Munich and Technical University of Munich) and Prof. Razansky (Eidgenösische Technische Hochschule Zurich) and is being further developed into a clinically applicable technology and sold commercially by the company iThera. As a first series of demonstrative clinical studies following rigorous technical development, MSOT will serve as a key tool for research partners in the investigation of several diseases that remain poorly-understood and have limited treatment options. These parallel studies will focus on lipedema and lymphedema as well as vascular malformations - three distinct disease groups with similarly unmet clinical needs for appropriate imaging modalities and high potential of translation to further major disease areas. By focusing on two unrelated diseases, this project will show the wide-reaching application of this innovative imaging approach. Following successful proof-of-principle validation in a clinical research environment, full exploitation and dissemination of the results will strive to deliver MSOT to the greater scientific community. The main objectives are to confirm/validate the spectral profile of fat and vasculature on MSOT in lipedema patients, to establish the spectral profile of vascular malformations based on MSOT for adults and children and to establish the spectral profile and imaging of lymphatic vessels.

With a detailed analysis of the architecture, our understanding of the physiology and pathology of the skin may be enhanced.

DETAILED DESCRIPTION:
To date, the diagnostic path of illnesses involving an altered adipose tissue architecture are usually slow and depend heavily on the experience of the examiner, so it often takes several years before the patient is properly treated. Current imaging methods for the quantitative assessment of subcutaneous fat tissue only provide non-specific findings. With our study, the investigators present a novel imaging method for examining adipose tissue.

Optoacoustics is an innovative hybrid imaging method that combines the high contrast of optical imaging with the high resolution of acoustics. The MSOT system used consists of a laser in the visible near-infrared and far-infrared wavelength range (660nm -1300nm) and an ultrasonic sensor connected to a computer. Using optical components, the area to be measured is illuminated with ultra-short light pulses of selectable wavelength. The light is absorbed to varying degrees inside the object - depending on the properties of the tissue. The Laser light stimulates chromophores such as hemoglobin or melanin in the human body, which results in an expansion and subsequent contraction of the tissue, the so-called thermoelastic effect. The local microscopic volume fluctuations emit pressure waves in the ultrasonic range (photoacoustic effect). The skin surface is scanned using high-precision microstages. At each location, the ultrasound signals generated by the light pulse are recorded tomographically outside the object using the detector and stored on the computer. With the help of special algorithms, the properties of the tissue can be reconstructed on the computer from the measured ultrasound signal. MSOT enables non-invasive, non-ionizing imaging with high spatial resolution (80 μm), which enables specific visualization of endogenous tissue pigments such as collagen fibers, fat, melanin, oxyhemoglobin and deoxyhemoglobin. Lasers for stimulating certain chromophores are already in wide therapeutic use in dermatology; their effects and side effects are known and are minimal to non-existent when a suitable energy is selected. The penetration depth of MSOT is significantly greater compared to other optical imaging methods.

In addition, this non-invasive, real-time measuring system can be used in numerous everyday clinical questions that otherwise require more invasive methods like CT or MRI. Apart from the examination of fatty tissue architecture, MSOT could be used pre- and perioperatively to visualize vessels, for example to optimize or even primarily enable the perfusion of flaps. The aim is to display and analyze the architecture of the subcutaneous fatty tissue in plastic surgery patients using MSOT.

The study is designed as a prospective cohort study of subjects recruited from the plastic surgery patient population. MSOT measurements are carried out on 50 subjects with clinically healthy subcutaneous fatty tissue and 50 subjects with changes in the subcutaneous fatty tissue (e.g. lipedema). The recorded data is quantified and compared.

The test subjects for this study are recruited from the trauma surgery, orthopedics and plastic surgery clinic and polyclinic. In particular, patients are recruited from the special plastic surgery consultation hours.

Everyone present wears laser safety goggles. An ultrasound gel film is applied to approximately 1 cm² of skin in several places on the selected extremities of the patient and the detector is placed on the gel film. These areas of skin are then scanned, with the areas to be examined being illuminated with ultra-short light pulses of a selectable wavelength. The resulting sound waves are detected with ultrasonic sensors and reconstructed on the computer and spectrally separated. A single measurement takes approximately 5 minutes. Including preparation, measuring the three skin areas will take approximately 20 minutes. Invasive procedures are not planned in this project.

The scanned areas are exported from the software as image material and stored pseudonymously. There is also photo documentation of the soft tissue that was scanned. These photos are also saved. To document health data, a lipedema documentation form is completed.

The optoacoustic modality does not require ionizing radiation and is based solely on the detection of acoustic waves induced by laser light. Both the technology of irradiation with various lasers and sonography are already widely used in the diagnosis and treatment of skin diseases. Therefore, their side effects are very predictable and, with appropriately selected energies, minimal to non-existent. To excite optoacoustic signals, class 4 pulsed lasers in the visible and near-infrared range (660 - 1300 nm) with a very short pulse duration (9ns) are used. The American National Standards Institute (ANSI) has set limit values for the use of lasers of this type, which are not exceeded in the experiments. Theoretically, treatment errors, such as choosing too high an energy level, can lead to tissue damage depending on the laser used. Lasers in the area of the chromophore hemoglobin can cause thermal vascular damage to the smallest and smallest vessels. If the energies are chosen to be very high, the maximum result could be local damage to the epidermis with subsequent local scarring, similar to a burn.

Since these effects are known through years of experience in widespread use, none of these side effects are expected during this study.

The evaluation of the sound waves generated using sonography is considered safe and no side effects are to be expected.

The laser light is directed onto the skin via the detector. Laser light can therefore only penetrate to the outside indirectly through scattering and theoretically reach the eyes of surrounding people. Since laser light with the above specification can be harmful to the eyes, care is taken to ensure that everyone present wears laser safety glasses during the measurement. There is virtually no risk of eye injury when wearing laser safety glasses.

The individual discontinuation criteria include intolerance and reactions such as redness. Previously described undesirable effects during treatment include redness and thermal vascular damage to soft tissue or subjectively perceived side effects. Another individual termination criterion is the revocation of the test subjects' consent to participate in the study or the refusal to wear laser safety glasses.

Termination criteria for the overall study include: unrecoverable defect in the monitoring system (MSOT), loss of all data. Redness with blistering in the sense of skin burns grade IIa (not yet described).

The aim of this pilot project is to describe the microarchitecture of the subcutaneous fatty tissue in patients with and without skin changes (e.g. lipedema) using MSOT. The ability to visualize these changes could lead to a better understanding of the physiology and pathophysiology of the skin.

When carrying out the investigation, the following guidelines and laws are observed:

* Declaration of Helsinki (2013) as supplemented by Venice 1983 and Hong Kong 1989
* The vote of the local ethics committee is obtained from the head of the scientific investigation
* The start and implementation of the investigation are tied to a vote by the ethics committee. After the investigation has been completed, a report or publication is submitted to the ethics committee
* The subjects' consent is given voluntarily after the risks have been explained. The test subjects do not receive any compensation
* Consent can be withdrawn at any time without giving reasons
* If the participant withdraws from the study, data material that has already been obtained will be destroyed or the subject will be asked whether he or she agrees to the evaluation of the material
* The names of the test subjects and all other confidential information are subject to medical confidentiality and the provisions of the Federal Data Protection Act (BDSG) - - Subject data may only be passed on in pseudonymized form. Third parties do not have access to the original documents
* Before the start of the study, the test subjects are informed in writing and orally about the nature and scope of the planned examinations, in particular about the possible benefits for their health and any risks. The participants consent is documented by signing the consent form

ELIGIBILITY:
Inclusion Criteria:

* Typical tenderness in the calf, back of the knee or lateral thigh
* Tendency to hematoma in areas affected by edema
* Typical inspection disorder of fatty tissue distribution with dent formation, asymmetry in lateral comparison and increased circumference
* Tendency to edema throughout the day with typical feeling of pressure/pain
* Unsuccessful conservative therapy attempts and weight loss attempts.

Exclusion Criteria:

* Age <18 or >80
* pregnancy and breastfeeding
* Lack of voluntary consent

Ages: 18 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: The subjects for this study are recruited from the trauma surgery, orthopedics and plastic surgery clinic and polyclinic. In particular, patients are recruited from the special plastic surgery consultation hours.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Visualization of subcutaneous fatty tissue | After inclusion of the subject the architecture of the subcutaneous fatty is visualized one time at baseline. There will be only one examination of each patient.
  The aim is to display and analyze the architecture of the subcutaneous fatty tissue in plastic surgery patients using MSOT

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsmedizin Göttingen, Göttingen, Lower Saxony, Germany